CLINICAL TRIAL: NCT02481245
Title: A Pan-PPAR Agonist Treatment for Bipolar Depression: A Proof of Concept Study
Brief Title: BezafibrateTreatment for Bipolar Depression: A Proof of Concept Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brain & Behavior Research Foundation (Other); J Willard and Alice S. Marriott Foundation (Unknown)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Director, Dauten Family Center for Bipolar Treatment Innovation, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000862
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Bipolar Disorder; Depressive Episode
Keywords: Bipolar Disorder; Bezafibrate; Depressive Episode
MeSH Terms: conditions — Bipolar Disorder | interventions — Bezafibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bipolar I and Bipolar II Disorder (Experimental): 30 currently depressed patients with DSM-IV bipolar I or bipolar II disorder who are currently taking an adequate dose of an FDA-approved anti-manic medication will receive Bezafibrate treatment.
  Interventions: Drug: Bezafibrate

INTERVENTIONS:
Drug: Bezafibrate — 30 patients with Bipolar I or Bipolar II disorder who are experiencing an acute bipolar depressive episode will be given bezafibrate XR 400 mg daily added on to adequate doses of an FDA-approved anti-manic medication.
  Other Names: Bezalip

SUMMARY:
We propose to test the hypothesis that bezafibrate, a pan-PPAR agonist, may be effective and safe for bipolar depression with the following specific aims:

Aim #1. Proof-of-Concept Safety and Tolerability Aim: To assess the safety and tolerability of bezafibrate added to anti-manic medication for bipolar depression, especially with regard to worsening manic symptoms and suicidal ideation.

We will conduct a phase IIa, 8-week, open pilot trial of bezafibrate added to FDA-approved anti-manic medication in 30 participants with bipolar depression. We will monitor changes in manic symptoms (Young Mania Rating Scale), suicidal ideation, cognitive functioning specifically in attention and verbal memory, and treatment emergent adverse events (SAFTEE). We will also monitor changes in the Framingham Cardiovascular Risk Score.

Aim #2. Preliminary Assessment of Efficacy: To assess the antidepressant efficacy of bezafibrate added to anti-manic medication for acute bipolar I major depressive episodes.

Hypothesis: The bezafibrate group will have a statistically significant decrease in the Montgomery Asberg Rating Scale (MADRS) Scores over 8 weeks. The results of this proof-of concept phase IIa study will help us to plan a placebo-controlled randomized trial. In summary, we propose an 8-week, proof-of-concept open pilot trial of an adjunctive pan-PPAR agonist, bezafibrate, for 30 patients with an acute bipolar I major depressive episode. The study may have a profound impact on the development of a novel treatment consistent with the mitochondrial dysregulation hypothesis of bipolar disorder and, to the best of our knowledge, will be the first proof-of-concept trial to assess a pan-PPAR agonist for bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between the ages of 18 and 65 (inclusive)
2. DSM IV diagnosis of Bipolar Disorder Type I or Bipolar Disorder Type II
3. Ability to sign the Informed Consent Form
4. Taking an adequate dose of any FDA-approved anti-manic medication for at least two weeks prior to enrollment
5. Agrees not to change medications during the study
6. Meets criteria for a current major depressive episode as defined and operationalized by the MINI and by a MADRS score of >18 at screen and baseline (randomization)
7. Does not meet criteria for current hypomanic or manic episode as defined and operationalized by the MINI

Exclusion Criteria:

1. The following DSM-IV diagnoses: (1) Bipolar NOS, (2) Cyclothymia, (3) Schizoaffective Disorder, (4) organic mental disorders, (5) substance use disorders, including alcohol, active within the 3 months, (6) schizophrenia, (7) delusional disorder, (8) psychotic disorders not elsewhere classified, (9) acute bereavement, (10) severe borderline or antisocial personality disorder, (11) OCD or OCD-spectrum disorders
2. Primary diagnosis of anxiety disorders or patients where the anxiety disorder is the primary focus of treatment
3. Patients with mood congruent or mood incongruent psychotic features
4. Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (e.g. oral contraceptives, intrauterine device, barrier methods, or total abstinence from intercourse; Depo Provera is acceptable if it is started 3 months prior to enrollment). Women who are nursing
5. Patients who are a serious suicide or homicide risk
6. Suspected or known clinically unstable systemic medical disorder including epilepsy, untreated endocrine disease, unstable angina, recent ulcers or significant esophagitis
7. Conditions which may be negatively affected by bezafibrate treatment, such as hepatobiliary disease
8. Clinical or laboratory evidence of hypothyroidism (if maintained on thyroid medication must be euthyroid for at least 1 month before Visit 1)
9. Subjects having failed two or more trials of somatic therapy (i.e., medications for bipolar depression or FDA-approved devices) during the current bipolar depressive episode
10. Current use of a fibrate or history of anaphylactic reaction or intolerance to fibrates or any component of the preparation
11. History of significant treatment non-adherence or situations where the subjects is unlikely to adhere to treatment, in the opinion of the investigator
12. History of stroke or cerebrovascular disease
13. Type 1 or Type II Diabetes requiring medication treatment treated with Pioglitazone or any other PPAR agonist medication.
14. Current use of of MAO Inhibitors, statins, and anticoagulants (e.g. warfarin)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 8 in Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline and Week 8
  The primary efficacy measure will be the change in MADRS score.

SECONDARY OUTCOMES:
Change from Baseline to Week 8 in Clinical Global Impressions Bipolar Scale (CGI-BP-S) score | Baseline and Week 8
  Secondary efficacy measure will be change in CGI-BP-S score.
Adiponectin Level at Baseline and Week 8 | Baseline and Week 8
  We will measure adiponectin as a well-established biomarker for the effect of bezafibrate on PPAR and examine changes in adiponectin as a mediator of changes in mood symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A. Nierenberg, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- The Dauten Family Center for Bipolar Treatment Innovation at Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Identifiable, individual-level data will not be shared. Deidentified group-level data will be published/presented after study completion and analysis.